CLINICAL TRIAL: NCT02984241
Title: EHealth Coping Skills Training for Women Whose Partner Has a Drinking Problem
Brief Title: E-Health Coping Skills Training for Women Whose Partner Has a Drinking Problem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: University of Oregon (Other)
Responsible Party: Principal Investigator, Robert Rychtarik, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AA024118
Record Dates: First submitted 2016-11-14; First posted 2016-12-06 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- eHealth Coping Skills Training + Coach (Active Comparator): Access to StopSpinningMyWheels.org + Coach Support
  Interventions: Behavioral: eHealth Coping Skills Training; Behavioral: Coach Support
- eHealth Coping Skills Training Only (Active Comparator): Access to StopSpinningMyWheels.org
  Interventions: Behavioral: eHealth Coping Skills Training
- eHealth Usual Web Care (Active Comparator): Access to StopSpinningMyWheels.org usual care
  Interventions: Behavioral: eHealth Usual Web Care

INTERVENTIONS:
Behavioral: eHealth Coping Skills Training — Access to a specialized coping skills training website
  Arms: eHealth Coping Skills Training + Coach; eHealth Coping Skills Training Only
Behavioral: eHealth Usual Web Care — Access to a website in which helpful information on coping that is available on the internet has been systematically collected and organized in one place for easy retrieval
  Arms: eHealth Usual Web Care
Behavioral: Coach Support — Access to a professional coach by phone
  Arms: eHealth Coping Skills Training + Coach

SUMMARY:
This study evaluates web-based interventions to help women cope with the stress arising from living with a problem-drinking partner

ELIGIBILITY:
Inclusion Criteria:

* Resides in New York State
* Fluent in English
* Male partner has an alcohol problem
* Computer access and smart phone
* Married or cohabiting

Exclusion Criteria:

* Substance use disorder
* Serious Mental Disorder
* Participation in prior studies
* Severe relationship violence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2019-10-13 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) Total Score | Change in BDI score up to 12 months postintervention
  A measure of depressive symptoms. Scores range from 0 to 63. Lower scores are indicative of better outcomes. A score of 14 or higher is considered clinically relevant.
State-Trait Anger Expression Inventory - 2 (STAXI-2, State Anger) | Change in STAXI score up to 12 months postintervention
  A measure of anger thoughts in their current state. Scores range from 1 to 60 with lower scores representing better outcomes. A score of 18 or above is considered clinically relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Rychtarik, Ph.D., Principal Investigator — University at Buffalo, Research Institute on Addictions; Brian G. Danaher, Ph.D., Principal Investigator — University of Oregon, Prevention Science Institute
Locations (1):
- Clinical and Research Institute on Addiction, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rychtarik RG, Danaher BG, McGillicuddy NB, Tyler MS, Barrick C, Leong F, Kosty DB. Web-Based Coping Skills Training and Coach Support for Women Living With a Partner With an Alcohol Use Disorder: Randomized Controlled Trial. J Med Internet Res. 2024 Aug 29;26:e56119. doi: 10.2196/56119. PMID 39208412